CLINICAL TRIAL: NCT01864824
Title: Air Pollution, Epigenetics and Cardiovascular Health: A Human Intervention Trial
Acronym: EPI-Air
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: University of Toronto (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Andrea Baccarelli, MD, PHD, MPH, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1R21ES021895-01 (NIH)
Record Dates: First submitted 2013-05-08; First posted 2013-05-30 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Heart Rate; Heart Rate Variability; Inflammation
Keywords: air pollution; particulate matter 2.5 (PM2.5); methyl donor; DNA methylation; mRNA; epigenetics; controlled human exposures; cardiovascular responses
MeSH Terms: conditions — Inflammation | interventions — Vitamin B 6; Vitamin B 12; Folic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methyl donor (Experimental): Methyl donor is made up of:
  2.5 mg of folic acid, 50 mg of vitamin B6, and 1 mg of vitamin B12 The design will include a 2 week placebo run-in followed by a baseline blank study (2-hrs exposure to medical air) to provide benchmarks for all assessed variables. Participants will then receive a 4-week placebo treatment before the first PM2.5 exposure study. A 4-week methyl-donor treatment (Dose: 2.5 mg of folic acid, 50 mg of vitamin B6, and 1 mg of vitamin B12 once a day) will precede the 2nd PM2.5 exposure.
  Interventions: Drug: methyl donor
- placebo (Placebo Comparator): placebo: The design will include a 2 week placebo run-in followed by a baseline blank study (2-hrs exposure to medical air) to provide benchmarks for all assessed variables. Participants will then receive a 4-week placebo treatment before the first PM2.5 exposure study. A 4-week methyl-donor treatment (Dose: 2.5 mg of folic acid, 50 mg of vitamin B6, and 1 mg of vitamin B12 once a day) will precede the 2nd PM2.5 exposure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methyl donor — The design will include a 2 week placebo run-in followed by a baseline blank study (2-hrs exposure to medical air) to provide benchmarks for all assessed variables. Participants will then receive a 4-week placebo treatment before the first PM2.5 exposure study. A 4-week methyl-donor treatment (Dose: 2.5 mg of folic acid, 50 mg of vitamin B6, and 1 mg of vitamin B12 once a day) will precede the 2nd PM2.5 exposure.
  Other Names: Vitamin B6; Vitamin B12; Folic Acid; Placebo
  Arms: methyl donor
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
In this study, the pills formulated are being used to try to ameliorate the effect of air pollution on epigenetic changes, specifically DNA methylation, potentially linked with particulate matter air pollution inhalation and cardiovascular health effects. The way in which this is achieved is that the vitamins, which act as methyl donors, add a methyl group to the DNA to reverse the loss observed on exposure to air pollution.

Specifically for this study, the methyl donor supplement has been made by Jamieson Laboratories, and consists of 50mg Vitamin B6 and 1 mg Vitamin B12, (both within Health Canada approved limits) and 2.5 mg folic acid. The non-vitamin ingredients are those commonly used in pill formation. However, the folic acid concentration is 2.5mg, which is above the 1.0mg limit set by Health Canada for a natural health product. This concentration, however, has been used in previous academic studies safely and effectively, and was also formulated by Jamieson Laboratories. (ClinicalTrials.gov number, NCT00106886; Current Controlled Trials number, ISRCTN14017017. HOPE2 study).

DETAILED DESCRIPTION:
Air pollution is a pervasive environmental threat estimated to cause ~800,000 deaths every year worldwide, mostly due to cardiovascular disease. This proposal addresses a fundamental mechanistic and pharmacologic question about effects of air pollution, which can most effectively be addressed through controlled human exposure experiments: does exposure have epigenetic effects that may have downstream subclinical or clinical consequences, and can adverse effects be safely reduced pharmacologically? Consistent evidence from in- vitro and human studies have shown that exposure to air particulate matter pollution (PM, i.e., fine particles) induces hypomethylation of the DNA, an epigenetic process that can underlie the activation of inflammatory genes and is postulated to link inhalation of PM into the lungs with cardiovascular inflammation and adverse responses. Our goal is to determine whether a pharmacological intervention with methyl-donors (i.e., folic acid, Vitamins B6 & B12, betaine, methionine, and choline) can avert this DNA methylation loss and mitigate the cardiovascular effects induced by PM exposure. The investigators will use experiments of human controlled exposure to PM - which reproduce conditions of exposure similar to those found in real life in urban environments - to conduct a double-blind, placebo-controlled crossover study. The investigators will test whether pharmacological intervention with methyl-donors attenuates the effects of PM exposure on DNA methylation (Aim 1), mRNA expression & plasma cytokines (Aim 2), and blood pressure, arterial vasoconstriction, endothelial function, and autonomic control of the heart (Aim 3). The investigators' study is poised to be the first human investigation to translate a wealth of animal data showing that methyl-donors can be used to modulate epigenetic states and avert environmental effects. The investigators have a unique opportunity to achieve this goal because we have access to one of the few facilities worldwide for human controlled-exposure studies, as well as to state-of-the-art resources for epigenetics investigations. The investigators will examine DNA methylation and mRNA expression in T-helper cells from human individuals, a cell type with key roles in determining adverse hypertensive and endothelial responses, as shown in several animal models. The investigators will test the effects of methyl-donors on a battery of cardiovascular endpoints that are highly sensitive to PM exposure. The investigators will explore the use of advanced statistical methods for mediation analyses to understand the relationships among PM, DNA methylation, RNA expression, plasma cytokines, and cardiovascular endpoints. The study will be conducted by an investigative team that has conducted seminal work in all of the research areas on which this proposal is built upon, including environmental epigenetics, cardiovascular effects of PM, and human controlled exposure studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age 18-60 years old
* Non-smoker
* must be able to fast 8 hours prior to exposure visits and for a further 4 hours during the exposure

Exclusion Criteria:

* Subjects must not be regularly taking multivitamins, vitamins C & E, folate, medications, fish oil or aspirin, oral or inhaled steroids, for 4 weeks before and during the trial.
* Lipid abnormalities
* Asthma or respiratory disease
* Hypertension (Bp> 140/90) or taking any blood pressure drug
* Known cardiac disease
* abnormal homocysteine or glucose levels

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
DNA methylation in circulating T-helper lymphocytes of six candidate genes (TNFa, TGFb, IFNg, IL17, IL2, IL6) | 2 years
  Blood will be collected from venous phlebotomy and processed for Th-cell isolation within 4hrs. DNA extraction will be performed manually on fresh unfrozen cells. DNA methylation analyses will be conducted using bisulfite-polymerase chain reaction-pyrosequencing. To select target sequences within each gene, we will rely both on assays from previous investigations and bioinformatic analysis using information from the genome browser on transcription factor binding sites conserved in the human/mouse/rat alignment, histone marks associated with active regulatory sequences and gene accessibility, and nucleosome occupancy. We will validate all assays using a titration curve of 0%-100% methylated DNA. Batch effect will be controlled by: a) using 0%, 50%, 100% methylation and universal DNA in each plate; b) running all samples from the same volunteer in one plate. We will intersperse 5% blind duplicates to test reproducibility. All samples will be assayed in duplicate runs.

SECONDARY OUTCOMES:
Blood pressure (BP) , brachial artery diameter (BAD), endothelium-dependent flow-mediated dilation (ED-FMD) and heart rate variability (HRV). | 2 years
  BP will be measured at 30-min intervals during exposure using an automated oscillometric ambulatory monitor secured on the upper left arm. Three BP measures will be taken at each time point separated by 1 minute, and the mean of the 2nd and 3rd measures used. BAD, FMD and nitroglycerin-mediated dilatation will be measured using a Terason 2000 ultrasound with a 7.5-10.0 megahertz linear array transducer. Peak FMD within this period will be used as our primary study outcome for endothelial function. Continuous EKG monitoring will be performed using high-resolution digital 12-lead Holter monitors. Holter monitoring will take place for 24-hr periods which will include before (pre-exposure testing), during the 2-hr exposure and post exposure (just after and 24-hrs post). Immediately prior to exposure, after the exposure and 24 hrs later, we will collect 10-minute resting supine HRV readings. HRV will be evaluated on 5-min ECG data using standardized techniques.

OTHER OUTCOMES:
mRNA expression of inflammatory genes (TNFa, TGFb, IFNg, IL17, IL2, IL6) in circulating T-helper lymphocytes; plasma cytokines. | 2 years
  We will extract total RNA from Th cells isolated and immediately preserved in mRNA later. We will design real-time PCR assays to measure mRNA levels of TNFα, IFNγ, IL-17, TGFβ, IL2 & IL6 following standardized procedures. All assays will be run in triplicates. We will measure 27 cytokines included in a pre-set Luminex Bio-Plex 27-plex panel. Analyses will include measures of the same mediators for which methylation analysis is measured (TNFα, IFNγ, IL-17, TGFβ, IL2, and IL6), which represent the strongest candidates for their roles in Th cells, as shown in cardiovascular models of hypertension. The remaining inflammatory mediators are IL7, IL8, IL12, GM-CSF, IL4, IL5, IL9, IL10, IL13, GM-CSF, IL1β, IL1ra, IL15, IL17, MCP1, MIP1α, MIP1β, PDGF-BB, VEGF, FGF, RANTES, IP-10, eotaxin, GCSF. Samples will be run in triplicates. Also, we will measure plasma CRP through a high-sensitivity method (Dade Behring).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Baccarelli, MD PHD MPH, Principal Investigator — HSPH; Frances Silverman, PHD, Study Director — Unity Health Toronto; Diane R. Gold, MD, Study Chair — HSPH
Locations (1):
- Gage Occupational and Environmental Health St. Michael's Hospital/University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Brook RD, Rajagopalan S, Pope CA 3rd, Brook JR, Bhatnagar A, Diez-Roux AV, Holguin F, Hong Y, Luepker RV, Mittleman MA, Peters A, Siscovick D, Smith SC Jr, Whitsel L, Kaufman JD; American Heart Association Council on Epidemiology and Prevention, Council on the Kidney in Cardiovascular Disease, and Council on Nutrition, Physical Activity and Metabolism. Particulate matter air pollution and cardiovascular disease: An update to the scientific statement from the American Heart Association. Circulation. 2010 Jun 1;121(21):2331-78. doi: 10.1161/CIR.0b013e3181dbece1. Epub 2010 May 10. PMID 20458016
- [Background] O'Toole TE, Conklin DJ, Bhatnagar A. Environmental risk factors for heart disease. Rev Environ Health. 2008 Jul-Sep;23(3):167-202. doi: 10.1515/reveh.2008.23.3.167. PMID 19119685
- [Background] Zanobetti A, Canner MJ, Stone PH, Schwartz J, Sher D, Eagan-Bengston E, Gates KA, Hartley LH, Suh H, Gold DR. Ambient pollution and blood pressure in cardiac rehabilitation patients. Circulation. 2004 Oct 12;110(15):2184-9. doi: 10.1161/01.CIR.0000143831.33243.D8. Epub 2004 Oct 4. PMID 15466639
- [Background] Brook RD, Rajagopalan S. Particulate matter, air pollution, and blood pressure. J Am Soc Hypertens. 2009 Sep-Oct;3(5):332-50. doi: 10.1016/j.jash.2009.08.005. PMID 20409976
- [Background] Brook RD, Bard RL, Burnett RT, Shin HH, Vette A, Croghan C, Phillips M, Rodes C, Thornburg J, Williams R. Differences in blood pressure and vascular responses associated with ambient fine particulate matter exposures measured at the personal versus community level. Occup Environ Med. 2011 Mar;68(3):224-30. doi: 10.1136/oem.2009.053991. Epub 2010 Oct 8. PMID 20935292
- [Background] Liu L, Ruddy T, Dalipaj M, Poon R, Szyszkowicz M, You H, Dales RE, Wheeler AJ. Effects of indoor, outdoor, and personal exposure to particulate air pollution on cardiovascular physiology and systemic mediators in seniors. J Occup Environ Med. 2009 Sep;51(9):1088-98. doi: 10.1097/JOM.0b013e3181b35144. PMID 19701101
- [Background] O'Neill MS, Veves A, Zanobetti A, Sarnat JA, Gold DR, Economides PA, Horton ES, Schwartz J. Diabetes enhances vulnerability to particulate air pollution-associated impairment in vascular reactivity and endothelial function. Circulation. 2005 Jun 7;111(22):2913-20. doi: 10.1161/CIRCULATIONAHA.104.517110. Epub 2005 May 31. PMID 15927967
- [Background] Baccarelli A, Cassano PA, Litonjua A, Park SK, Suh H, Sparrow D, Vokonas P, Schwartz J. Cardiac autonomic dysfunction: effects from particulate air pollution and protection by dietary methyl nutrients and metabolic polymorphisms. Circulation. 2008 Apr 8;117(14):1802-9. doi: 10.1161/CIRCULATIONAHA.107.726067. Epub 2008 Mar 31. PMID 18378616
- [Background] Adar SD, Gold DR, Coull BA, Schwartz J, Stone PH, Suh H. Focused exposures to airborne traffic particles and heart rate variability in the elderly. Epidemiology. 2007 Jan;18(1):95-103. doi: 10.1097/01.ede.0000249409.81050.46. PMID 17149139
- [Result] Zhong J, Trevisi L, Urch B, Lin X, Speck M, Coull BA, Liss G, Thompson A, Wu S, Wilson A, Koutrakis P, Silverman F, Gold DR, Baccarelli AA. B-vitamin Supplementation Mitigates Effects of Fine Particles on Cardiac Autonomic Dysfunction and Inflammation: A Pilot Human Intervention Trial. Sci Rep. 2017 Apr 3;7:45322. doi: 10.1038/srep45322. PMID 28367952
- [Result] Zhong J, Karlsson O, Wang G, Li J, Guo Y, Lin X, Zemplenyi M, Sanchez-Guerra M, Trevisi L, Urch B, Speck M, Liang L, Coull BA, Koutrakis P, Silverman F, Gold DR, Wu T, Baccarelli AA. B vitamins attenuate the epigenetic effects of ambient fine particles in a pilot human intervention trial. Proc Natl Acad Sci U S A. 2017 Mar 28;114(13):3503-3508. doi: 10.1073/pnas.1618545114. Epub 2017 Mar 13. PMID 28289216
- [Result] Zhong J, Urch B, Speck M, Coull BA, Koutrakis P, Thorne PS, Scott J, Liu L, Brook RD, Behbod B, Gibson H, Silverman F, Mittleman MA, Baccarelli AA, Gold DR. Endotoxin and beta-1,3-d-Glucan in Concentrated Ambient Particles Induce Rapid Increase in Blood Pressure in Controlled Human Exposures. Hypertension. 2015 Sep;66(3):509-16. doi: 10.1161/HYPERTENSIONAHA.115.05342. Epub 2015 Jun 29. PMID 26123683